CLINICAL TRIAL: NCT00591409
Title: A Multi-Center, Randomized, Open-Label, Prospective Bridging, Parallel Dose-Finding Trial Comparing Efficacy, Safety and Pharmacokinetics of 4 Doses of Org 25969 and Placebo Administered at Reappearance of T2 After Rocuronium or Vecuronium in Japanese and Caucasian Subjects. Part A: Japanese Subjects
Brief Title: A Bridging Trial Comparing Sugammadex (Org 25969) at Reappearance of T2 in Japanese and Caucasian Participants. Part A: Japanese Participants (P05956)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05956; 19.4.208A (Other: Organon Protocol Number); MK-8616-030 (Other: Merck Protocol Number)
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Rocuronium + Placebo (Placebo Comparator): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered intravenously (IV), followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of T2 a single dose of placebo was administered IV.
  Interventions: Drug: Placebo
- Rocuronium + 0.5 mg/kg sugammadex (Experimental): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered IV, followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of T2 a single dose of 0.5 mg/kg sugammadex was administered IV.
  Interventions: Drug: sugammadex
- Rocuronium + 1.0 mg/kg sugammadex (Experimental): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered IV, followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of T2 a single dose of 1.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: sugammadex
- Rocuronium + 2.0 mg/kg sugammadex (Experimental): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered IV, followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of T2 a single dose of 2.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: sugammadex
- Rocuronium + 4.0 mg/kg sugammadex (Experimental): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered IV, followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of T2 a single dose of 4.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: sugammadex
- Vecuronium + Placebo (Placebo Comparator): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.04 mg/kg vecuronium IV if necessary. At reappearance of T2 a single dose of placebo was administered IV.
  Interventions: Drug: Placebo
- Vecuronium + 0.5 mg/kg sugammadex (Experimental): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.04 mg/kg vecuronium IV if necessary. At reappearance of T2 a single dose of 0.5 mg/kg sugammadex was administered IV.
  Interventions: Drug: sugammadex
- Vecuronium + 1.0 mg/kg sugammadex (Experimental): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.04 mg/kg vecuronium IV if necessary. At reappearance of T2 a single dose of 1.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: sugammadex
- Vecuronium + 2.0 mg/kg sugammadex (Experimental): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.04 mg/kg vecuronium IV if necessary. At reappearance of T2 a single dose of 2.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: sugammadex
- Vecuronium + 4.0 mg/kg sugammadex (Experimental): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.04 mg/kg vecuronium IV if necessary. At reappearance of T2 a single dose of 4.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: sugammadex

INTERVENTIONS:
Drug: sugammadex — After induction of anesthesia an intubation dose of NMBA was administered IV: either 0.9 mg/kg rocuronium or 0.1 mg/kg vecuronium.
  Maintenance doses of 0.1-0.2 mg/kg rocuronium IV or 0.02-0.04 mg/kg vecuronium IV could be administered if necessary.
  At reappearance of T2 the randomized single dose of sugammadex (0.5 to 4 mg/kg) IV was administered.
  Other Names: Org 25969
  Arms: Rocuronium + 0.5 mg/kg sugammadex; Rocuronium + 1.0 mg/kg sugammadex; Rocuronium + 2.0 mg/kg sugammadex; Rocuronium + 4.0 mg/kg sugammadex; Vecuronium + 0.5 mg/kg sugammadex; Vecuronium + 1.0 mg/kg sugammadex; Vecuronium + 2.0 mg/kg sugammadex; Vecuronium + 4.0 mg/kg sugammadex
Drug: Placebo — After induction of anesthesia an intubation dose of NMBA was administered IV: either 0.9 mg/kg rocuronium or 0.1 mg/kg vecuronium.
  Maintenance doses of 0.1-0.2 mg/kg rocuronium IV or 0.02-0.04 mg/kg vecuronium IV could be administered if necessary.
  At reappearance of T2 the randomized single dose of placebo IV was administered
  Arms: Rocuronium + Placebo; Vecuronium + Placebo

SUMMARY:
The objective of this trial was to establish the dose-response of T2 (the amplitude of the first response of second twitch to train of four (TOF) stimulation, expressed as percentage of control first twitch,T1) in Japanese and Caucasian participants. Part A: Japanese Participants

DETAILED DESCRIPTION:
For most surgical procedures a depth of neuromuscular block of 1-2 twitches after TOF-stimulation is sufficient to avoid unwanted muscular activity. At reappearance of T2, the anesthesiologist might decide to either give (another) maintenance dose of rocuronium or vecuronium when surgery continues, to await spontaneous recovery of neuromuscular block or to reverse the neuromuscular block. Sugammadex (Org 25969) has been shown in previous trials to greatly reduce the time to full recovery when administered at reappearance of T2, both after rocuronium- and vecuronium-induced neuromuscular blockade. The current trial P05956 was conducted in Japan and set up to establish the dose-response relationship of sugammadex given during sevoflurane anesthesia at reappearance of T2 after rocuronium or vecuronium in Japanese participants. In addition to recovery time, also pharmacokinetics and safety of sugammadex were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Is of American Society of Anesthesiologists (ASA) class 1 - 3;
* Is at least 20 years but under 65 years of age;
* Japanese participants;
* Is scheduled for elective surgery in supine position and under sevoflurane anesthesia, in need of administration of neuromuscular blocking agents (NMBAs), with an anticipated duration of about 1.5-3 hours;
* Has given written informed consent.

Exclusion Criteria:

* Participants in whom a difficult intubation because of anatomical malformations was expected;
* Is known or suspected to have neuromuscular disorders impairing the effect of NMBAs and/or significant renal dysfunction (for example a creatinine level > 1.6 mg/dl) and/or severe hepatic dysfunction.
* Is known or suspected to have a (family) history of malignant hyperthermia;
* Is known or suspected to have an allergy to narcotics, muscle relaxants or other medication used during general anesthesia;
* Is receiving medication expected to interfere with the rocuronium or vecuronium given in this trial, based on the dose and time of administration;
* Females who were pregnant;
* Females not using birth control or using only oral contraception as birth control continuously;
* Were breast-feeding;
* Has already participated in P05956, or in another trial with sugammadex;
* Has participated in another clinical trial within 6 months of entering into P05956

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-01-03 (Actual); Primary Completion 2006-09-22 (Actual); Study Completion 2006-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Takeda J, Iwasaki H, Yamakage M, Ozaki M, Kawamata M, Hatano Y, Yorozuya T, Miyakawa H, Kanmura Y. [Efficacy and safety of sugammadex (Org 25969) in reversing moderate neuromuscular block induced by rocuronium or vecuronium in Japanese patients]. Masui. 2014 Oct;63(10):1075-82. Japanese. PMID 25693332
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Japanese participants who had a surgical procedure using a general anesthesia of rocuronium or vecuronium for endotracheal intubation and maintenance of neuromuscular block were enrolled in this study.
Period: Overall Study
Arm/Group | Rocuronium + Placebo | Rocuronium + 0.5 mg/kg Sugammadex | Rocuronium + 1.0 mg/kg Sugammadex | Rocuronium + 2.0 mg/kg Sugammadex | Rocuronium + 4.0 mg/kg Sugammadex | Vecuronium + Placebo | Vecuronium + 0.5 mg/kg Sugammadex | Vecuronium + 1.0 mg/kg Sugammadex | Vecuronium + 2.0 mg/kg Sugammadex | Vecuronium + 4.0 mg/kg Sugammadex
Started | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 9 | 11
Treated | 10 | 10 | 10 | 10 | 9 | 10 | 10 | 10 | 9 | 10
Completed | 10 | 10 | 10 | 10 | 9 | 10 | 10 | 10 | 9 | 10
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Not Treated | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All Participants As Treated
Groups:
- Rocuronium + Placebo: After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered IV, followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of T2 a single dose of placebo was administered IV.
- Total: Total of all reporting groups
Arm/Group | Rocuronium + Placebo | Rocuronium + 0.5 mg/kg Sugammadex | Rocuronium + 1.0 mg/kg Sugammadex | Rocuronium + 2.0 mg/kg Sugammadex | Rocuronium + 4.0 mg/kg Sugammadex | Vecuronium + Placebo | Vecuronium + 0.5 mg/kg Sugammadex | Vecuronium + 1.0 mg/kg Sugammadex | Vecuronium + 2.0 mg/kg Sugammadex | Vecuronium + 4.0 mg/kg Sugammadex | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 9 | 10 | 10 | 10 | 9 | 10 | 98
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41 (10) | 44 (10) | 49 (9) | 45 (10) | 41 (15) | 49 (14) | 49 (8) | 46 (13) | 52 (13) | 44 (14) | 46 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 5 | 5 | 7 | 6 | 5 | 6 | 5 | 3 | 54
  Male | 5 | 3 | 5 | 5 | 2 | 4 | 5 | 4 | 4 | 7 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 10 | 10 | 9 | 10 | 10 | 10 | 9 | 10 | 98
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time From Start of Administration of Sugammadex or Placebo to Recovery of the Fourth Twitch/First Twitch (T4/T1) Ratio to 0.9
Description: Neuromuscular functioning was monitored by applying repetitive Train-Of-Four (TOF) electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the amplitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from neuromuscular blockade (NMB). In this study, twitch responses were recorded until the T4/T1 Ratio reached >= 0.9, the minimum acceptable ratio that indicated recovery from NMB. A faster time to recovery of the T4/T1 Ratio to 0.9 indicates a faster recovery from NMB.
Time Frame: Day 1: From start of sugammadex or placebo administration to recovery of T4/T1 ratio to 0.9 (up to 24 hours)
Population: All randomized participants who received sugammadex or placebo; without any protocol violations, and who had at least one post baseline efficacy measurement, who had a TOF trace, had a reliable TOF trace, and where drug administration did not interfere with the effect of rocuronium or vecuronium.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Rocuronium + Placebo | Rocuronium + 0.5 mg/kg Sugammadex | Rocuronium + 1.0 mg/kg Sugammadex | Rocuronium + 2.0 mg/kg Sugammadex | Rocuronium + 4.0 mg/kg Sugammadex | Vecuronium + Placebo | Vecuronium + 0.5 mg/kg Sugammadex | Vecuronium + 1.0 mg/kg Sugammadex | Vecuronium + 2.0 mg/kg Sugammadex | Vecuronium + 4.0 mg/kg Sugammadex
Number analyzed (Participants) | 6 | 5 | 10 | 7 | 9 | 7 | 3 | 8 | 6 | 10
Minutes | 82.08 (27.57) | 3.95 (2.50) | 2.48 (1.28) | 2.17 (1.23) | 1.85 (1.17) | 83.20 (20.63) | 52.03 (64.92) | 10.63 (19.23) | 2.77 (0.83) | 2.08 (0.90)

2. Secondary Outcome: Time From Start of Administration of Sugammadex or Placebo to Recovery of the T4/T1 Ratio to 0.7
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the amplitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB. A faster time to recovery of the T4/T1 Ratio to 0.7 indicates a faster recovery from NMB.
Time Frame: Day 1: From start of sugammadex or placebo administration to recovery of T4/T1 ratio to 0.7 (up to 24 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Rocuronium + Placebo | Rocuronium + 0.5 mg/kg Sugammadex | Rocuronium + 1.0 mg/kg Sugammadex | Rocuronium + 2.0 mg/kg Sugammadex | Rocuronium + 4.0 mg/kg Sugammadex | Vecuronium + Placebo | Vecuronium + 0.5 mg/kg Sugammadex | Vecuronium + 1.0 mg/kg Sugammadex | Vecuronium + 2.0 mg/kg Sugammadex | Vecuronium + 4.0 mg/kg Sugammadex
Number analyzed (Participants) | 7 | 5 | 10 | 9 | 9 | 9 | 4 | 9 | 8 | 10
Minutes | 52.60 (16.27) | 2.35 (0.70) | 1.73 (0.85) | 1.23 (0.38) | 1.20 (0.27) | 85.85 (75.12) | 12.52 (17.95) | 2.87 (1.13) | 2.30 (0.60) | 1.33 (0.43)

3. Secondary Outcome: Time From Start of Administration of Sugammadex or Placebo to Recovery of the T4/T1 Ratio to 0.8
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the amplitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB. A faster time to recovery of the T4/T1 Ratio to 0.8 indicates a faster recovery from NMB.
Time Frame: Day 1: From start of sugammadex or placebo administration to recovery of T4/T1 ratio to 0.8 (up to 24 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Rocuronium + Placebo | Rocuronium + 0.5 mg/kg Sugammadex | Rocuronium + 1.0 mg/kg Sugammadex | Rocuronium + 2.0 mg/kg Sugammadex | Rocuronium + 4.0 mg/kg Sugammadex | Vecuronium + Placebo | Vecuronium + 0.5 mg/kg Sugammadex | Vecuronium + 1.0 mg/kg Sugammadex | Vecuronium + 2.0 mg/kg Sugammadex | Vecuronium + 4.0 mg/kg Sugammadex
Number analyzed (Participants) | 6 | 5 | 10 | 9 | 9 | 7 | 3 | 9 | 8 | 10
Minutes | 63.67 (21.77) | 2.70 (1.00) | 1.87 (0.98) | 1.50 (0.55) | 1.32 (0.35) | 68.40 (19.58) | 5.55 (1.90) | 3.75 (1.45) | 3.08 (1.68) | 1.63 (0.48)

ADVERSE EVENTS:
Time Frame: Up to 7 days after sugammadex or placebo treatment
Description: All participants as treated
Arm/Group | Rocuronium + Placebo | Rocuronium + 0.5 mg/kg Sugammadex | Rocuronium + 1.0 mg/kg Sugammadex | Rocuronium + 2.0 mg/kg Sugammadex | Rocuronium + 4.0 mg/kg Sugammadex | Vecuronium + Placebo | Vecuronium + 0.5 mg/kg Sugammadex | Vecuronium + 1.0 mg/kg Sugammadex | Vecuronium + 2.0 mg/kg Sugammadex | Vecuronium + 4.0 mg/kg Sugammadex
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/9 | 0/10 | 0/10 | 0/10 | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 1/10 | 0/9 | 0/10 | 1/10 | 0/10 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 10/10 | 9/10 | 8/9 | 10/10 | 9/10 | 9/10 | 9/9 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rocuronium + Placebo (N=10) | Rocuronium + 0.5 mg/kg Sugammadex (N=10) | Rocuronium + 1.0 mg/kg Sugammadex (N=10) | Rocuronium + 2.0 mg/kg Sugammadex (N=10) | Rocuronium + 4.0 mg/kg Sugammadex (N=9) | Vecuronium + Placebo (N=10) | Vecuronium + 0.5 mg/kg Sugammadex (N=10) | Vecuronium + 1.0 mg/kg Sugammadex (N=10) | Vecuronium + 2.0 mg/kg Sugammadex (N=9) | Vecuronium + 4.0 mg/kg Sugammadex (N=10)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intrauterine infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rocuronium + Placebo (N=10) | Rocuronium + 0.5 mg/kg Sugammadex (N=10) | Rocuronium + 1.0 mg/kg Sugammadex (N=10) | Rocuronium + 2.0 mg/kg Sugammadex (N=10) | Rocuronium + 4.0 mg/kg Sugammadex (N=9) | Vecuronium + Placebo (N=10) | Vecuronium + 0.5 mg/kg Sugammadex (N=10) | Vecuronium + 1.0 mg/kg Sugammadex (N=10) | Vecuronium + 2.0 mg/kg Sugammadex (N=9) | Vecuronium + 4.0 mg/kg Sugammadex (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 4 (4) | 4 (4) | 4 (4) | 4 (4) | 5 (6) | 4 (5) | 5 (5) | 1 (1)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palatal oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 3 (3) | 2 (2) | 0 (0)
Application site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Instillation site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Instillation site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower extremity mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral coldness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Puncture site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 3 (3) | 5 (5) | 3 (3) | 3 (3) | 5 (5) | 4 (4) | 2 (2) | 4 (4) | 2 (2)
Thirst (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venipuncture site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaesthetic complication cardiac (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Mental status changes postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural oedema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 4 (6) | 2 (2) | 1 (1) | 2 (3) | 1 (1) | 2 (2)
Procedural hypertension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 8 (8) | 7 (7) | 7 (7) | 6 (7) | 8 (8) | 9 (9) | 7 (7) | 9 (9) | 5 (5) | 8 (8)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Albumin urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Beta 2 microglobulin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Beta 2 microglobulin urine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body temperature decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Red blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Intracranial hypotension (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigeminal palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Tension (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital pruritus female (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulval erythema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngolaryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any scientific paper, presentation, or other communication concerning this clinical trial will first be submitted to the Sponsor, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.